CLINICAL TRIAL: NCT05509738
Title: Feasibility of A Text Message-Based Healthcare Assistant in Pediatric Lower Urinary Tract Symptoms Care
Brief Title: Feasibility of Text4US Program
Acronym: Text4US
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Recruitment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kathleen Kan, CLINICAL ASSISTANT PROFESSOR, UROLOGY, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 65815
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Reminder Systems; Text Messaging; Urinary Dysfunction; Urinary Bladder; Behavior Change Techniques

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two groups that differ only in the order of receiving the text message-based healthcare assistance as an adjunct to their children's standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Diaries - SMS (Experimental): Group 1 will be asked to complete a 2-day bladder diary + food diary during the first two weeks of the study, then will receive SMS Text reminders during the last 2 weeks of the study.
  Both groups will complete a pre-survey at the beginning of the study and a post-survey after each phase of the study (total 2 post-surveys).
  Interventions: Behavioral: SMS Text Messaging
- Group 2: SMS - Diaries (Experimental): Group 2 will receive SMS Text reminders during the first 2 weeks of the study, and then will be asked to complete a 2-day bladder diary + food diary during the last two weeks of the study.
  Both groups will complete a pre-survey at the beginning of the study and a post-survey after each phase of the study (total 2 post-surveys).
  Interventions: Behavioral: SMS Text Messaging

INTERVENTIONS:
Behavioral: SMS Text Messaging — The text message-based healthcare assistance includes 1) message reminders and 2) a daily achievement reflection. The delivery schedule is as below.
  1. Message reminders:
     The investigators will send participants two text reminders per day, one in the morning and one in the afternoon, from Monday to Friday, with the information on helping their child achieve healthy bladder goals.
  2. Daily achievement reflection:
  The investigators will send participants a text message with a survey link to reflect their and their children's daily goal achievement Monday to Friday evenings. Timely feedback (e.g., inspirational and compliment messages) will be provided based on participants' responses.

SUMMARY:
Pediatric Lower Urinary Tract Symptoms (pLUTS) is common in school-age children and can negatively impact the quality of their life. Although at least 50% of children with pLUTS can improve through behavioral changes, how to support parents in helping their children adopt healthy bladder behaviors remains unrevealed. To solve this problem, the investigators developed an early model of a text message-based healthcare assistant. The aim of this study is to examine the feasibility of the text message-based healthcare assistant in pLUTS care.

DETAILED DESCRIPTION:
In this study, an early model of a text message-based healthcare assistant will be configured. The service provided by the proposed healthcare assistant includes (1) daily message reminders, and (2) daily achievement reflection. By employing the text message-based healthcare assistant in pLUTS care, the investigators hope to learn:

1. If the text message-based healthcare assistant could support parents of children with pLUTS in helping their children adopt healthy bladder behaviors?
2. What is parents' experience with the text message-based healthcare assistant in pLUTS care?
3. How to improve the text-message-based healthcare assistant in the future?

To date, these questions have not been answered in the existing literature on digital health. The study findings will deepen the understanding of treatment options for pLUTS and provide an opportunity to optimize pediatric urology practice by integrating digital technology.

The study aims to evaluate the feasibility of using a text message-based healthcare assistant to support parents of children with LUTS in helping their children adopt healthy bladder behaviors. Therefore, the involvement of human subjects is necessary.

Parents/guardians of children (5-18 years old) who present to the pediatric urology outpatient clinic for the first visit for pLUTS or attend a clinic program called Bladder Bootcamp (a one-hour Zoom urotherapy education session in a non-medical, group setting) will be identified. Clinic staff or Bladder Bootcamp instructors will introduce the research staff to potential participants during the waiting time. A research team member will neutrally invite potential participants to participate in the study by briefly describing it. For those who are not interested, the research team member will thank them for their time and not proceed forward. For those who are interested, the research team member will provide them with further study details, screen their eligibility, and review the consent form with those who are eligible. The consent form will emphasize that:

1. participation is voluntary.
2. participation will not affect the care under any circumstances.
3. participants can end participation at any time.
4. research staff will never share participants' identities with anyone else (confidentiality will be maintained).

Upon taking the consent, the study will be conducted. The total length of the study is four weeks. Participants will spend two weeks using a bladder diary and food diary to record their child's behaviors for 2 days (a part of standard care). They will spend another two weeks receiving personalized healthcare assistance via text messaging as an adjunct to their child's standard care. The order of using bladder and food diaries and receiving test messages-based healthcare assistance depends on which group participants were randomly assigned. The purpose of randomly assigning participants into two groups is to reduce research biases.

Specifically, the study has three phases:

Phase I: At the beginning of the study

* Evaluate participants' ability to receive text messages
* Provide participants with all the materials they need for this study, including bladder diary, food diary, participants instruction, and a bladder health education handout.
* Use an online survey to collect participants' and their child's basic information (e.g., demographic data, phone usage)

Phase II: During the 2 weeks of using bladder and food diaries

* Ask participants to fill out a bladder diary and food diary for 2 days
* Send participants an online survey asking about their experience with the bladder and food diaries

Phase III: During the 2 weeks of receiving text messages

* Provide participants the text message-based healthcare assistance.
* Send participants an online survey asking about their experience with the text message-based healthcare assistant.

The text message-based healthcare assistance provided in Phase III includes 1) message reminders and 2) a daily achievement reflection. The delivery schedule is as below. The delivery schedule is as below.

1. Message reminders:

   The investigators will send participants two text reminders per day, one in the morning and one in the afternoon, from Monday to Friday, with the information on helping their child achieve healthy bladder goals.
2. Daily achievement reflection:

The investigators will send participants a text message with a survey link to reflect their and their children's daily goal achievement Monday to Friday evenings. Timely feedback (e.g., inspirational and compliment messages) will be provided based on participants' responses.

To increase the response rate, Phase I will be conducted after taking the consent and in the presence of the research team member. For participants recruited in the clinic, they will fill out the survey using the university encrypted devices (e.g., research iPad) provided by the research team member (e.g., research iPad). If participants prefer to fill out the survey using their own devices, the research team member will send the survey link to them. For participants recruited in Bladder Bootcamp (online recruitment), they need to fill out the survey using the survey link provided by the research team member.

Given that participants may not complete all the surveys or answer all the questions in the survey, missing data may exist. If participants drop out from the study, the investigators will recruit another participant to replace the one who dropped out. The data of the person who dropped out will be destroyed.

All study-related materials (e.g., surveys, text messages, bladder and food diaries) have been attached to Section 16 of the protocol. The investigators may use a shortened version of the text messages for the study. If there are any changes to the study-related materials, the investigators will revise the IRB and upload the final materials.

All text messages (including survey links sent via text messages) will be encrypted and sent by RedCap by using a third-party web service named Twilio, which announces HIPAA eligibility in SMS. Participants' responses will be directly entered into RedCap and will not be collected and stored in Twilio.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians (above the age of 18) of children (5-18 years old) who have completed potty training with pLUTS.
* Parents/patients that have never completed a bladder/food diary before
* Fluent in English
* Able to receive text messages on a mobile device
* Referred with a diagnosis of LUTS in our outpatient clinic

Exclusion Criteria:

1. Parents/guardians of children with

   1. neurogenic bladder
   2. Genitourinary (GU) abnormalities
   3. Detrusor sphincter dyssynergia (DSD)
   4. renal transplant patients (pre and post)
   5. abdominal or spinal surgeries within one year
   6. other chronic illness that is known to affect LUTS
   7. currently on immunosuppression of any kind
   8. younger than 5 years old or older than 18 years old
2. Younger than 18 years old
3. Not fluent in English
4. Not able to receive text messages
5. filled out a bladder and/or food diary before

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Text-Messaging System | 3 years
  The feasibility of the Text4US program as assessed by:
  1. study recruitment and retention rates
  2. time required to recruit target participants
  3. cost associated with developing the Text4US program and maintaining the program until the completion of data collection
  4. participants' mobile/cell phone usage and preferred healthcare tools (assessed in pre-survey)
  5. differences in completion rates between bladder and food diaries (control condition) and reflection surveys (intervention condition).
Usefulness and Acceptability of the Text4US program | 3 years
  The usefulness and acceptability of the Text4US program as assessed by post-surveys adapted from Agyapong et al. (2013) with questions focusing on participants' engagement, satisfaction, experience, and intention to use. The responses differences between post-surveys of bladder and food diaries (control condition) and the Text4US program (intervention condition) will be examined. Besides, open-ended questions in post-surveys asking for participants' suggestions about the Text4US program will also be qualitatively analyzed.
Effectiveness of the Text4US program | 3 years
  The effectiveness of the Text4US program as assessed by:
  1. participants' self-efficacy: one 5-point Likert Scale question focusing on participants' self-efficacy in healthy bladder behavior adoption, changes from baseline to the end of bladder & food diaries phase (control condition), and the end of the Text4US phase (intervention condition)
  2. participants' perceived effects: differences in participants' perceived effects of bladder and food diaries (control condition) and the Test4US program (intervention condition) on bladder health. Assessment questions are adapted from Agyapong et al. (2013) and presented in post-surveys.
  3. children's healthy bladder behavior: differences in participant's self-reported healthy bladder behavior between bladder and food diaries (control condition) and reflection surveys (intervention condition).

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Identifiers might be removed from identifiable private information and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies. Any shared data will be de-identified.